CLINICAL TRIAL: NCT03495375
Title: Randomized Placebo-controlled Treatment of Impulsivity in Adults With Probiotics
Brief Title: Treating Impulsivity in Adults With Probiotics
Acronym: PROBIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Vall d'Hebron (Other)
Collaborators: Goethe University (Other); Semmelweis University (Other); University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Josep Antoni Ramos-Quiroga, Head of Department of Psychiatry, Hospital Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HValldhebron
Record Dates: First submitted 2018-02-26; First posted 2018-04-12 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Impulsive Behavior; Compulsive Disorder; ADHD; Borderline Personality Disorder
Keywords: Impulsivity; Compulsivity; Aggression; Microbiome; Probiotic; Nutrition; Psychiatric disorders; Synbiotic2000Forte
MeSH Terms: conditions — Impulsive Behavior; Compulsive Personality Disorder; Attention Deficit Disorder with Hyperactivity; Borderline Personality Disorder; Aggression; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with a probiotic (Experimental): Synbiotic2000Forte (SF) it is composed of 3 LAB species known to have anti-inflammatory effects and restoring the intestinal barrier, and 4 fermentable fibers: Pediococcus pentosaceus 5-33:3, Lactobacillus paracasei subsp paracasei 19, and Lactobacillus plantarum 2362 in combination with the following four fermentable fibres: betaglucan, inulin, pectin and resistant starch, a formula that is currently produced by Synbiotic AB, Sweden.
  Interventions: Dietary Supplement: Treatment with a probiotic
- Treatment with placebo powder (Placebo Comparator): Placebo will be a non-digestable carbohydrate with similar texture and flavor to the SF also provided by Synbiotic AB, Sweden.
  Interventions: Other: Treatment with placebo

INTERVENTIONS:
Dietary Supplement: Treatment with a probiotic — All participants will take the probiotic once daily for 10 weeks in the form of a powder that can be spread on top of cold foods such as muesli, salad, or yogurt.
  Arms: Treatment with a probiotic
Other: Treatment with placebo — All participants will take the placebo once daily for 10 weeks.
  Arms: Treatment with placebo powder

SUMMARY:
A multicentre randomized double-blind placebo controlled parallel design (10 weeks) study investigating probiotic supplementation in highly impulsive adults (18-65 yrs; N=180). The probiotic studied is Synbiotic2000Forte that contain three well-studied anti-inflammatory lactic acid bacteria (LABs) and four fermentable fibers: Pediococcus pentosaceus 5-33:3, Lactobacillus paracasei subsp paracasei 19, and Lactobacillus plantarum 2362 in combination with the following four fermentable fibres: betaglucan, inulin, pectin and resistant starch. With this study we aim to detect, whether treatment with probiotics is effective in adults with high levels of impulsivity, compulsivity, and aggression.

DETAILED DESCRIPTION:
Impulsivity is a cross-disorder trait relevant in several psychiatric disorders, e.g. Attention Deficit Hyperactivity Disorder (ADHD) and Borderline Personality Disorder (BPD). They place a significant burden on patients, families and society in general. Only adults (aged 18 - 65 years) with a diagnosis of ADHD and/or BPD will be included in this study. We will also try to include at least 30% female participants to gender-balance the study.

Recruitment and treatment of participants will be provided at three trial centres: Vall d'Hebron Research Institute (VHIR), Goethe University Frankfurt (GU), Semmelweis University (SU), each enrolling 60 participants. Randomization to receive either Synbiotic2000Forte or placebo will be performed when signed informed assent by the participant has been obtained, eligibility checks have been conducted and at baseline assessment. An independent randomization service (www.randomization.com) will be used to ensure reliability and credibility in the randomization process. The study is double-blinded; neither the participants nor the clinicians involved in the study will have access to the randomization list.

In this placebo-controlled 10-week, we will evaluate a probiotic formula for oral administration called Synbiotic2000Forte (SF). Participants will take the probiotic once daily in the form of a powder that can be spread on top of cold foods such as muesli, salad, or yoghurt. Placebo will be a non-digestable carbohydrate with similar texture and flavor to the SF. Participants will be assessed at baseline before treatment is started (baseline demographics and primary- and secondary outcome measures will be collected and then monitored every five weeks for a total of 5 visits.

Proper conduct of data collection in the trial will be monitored by on-site visits of a monitoring staff throughout the study, and quality of data collected will further be monitored regularly by a statistical supervision team. Questionnaire data will be collected through Castor. All information collected in this study will remain strictly confidential. Data of participants will be coded in such a way that participants cannot be identified from the corresponding data according to the regulations (unique pseudocode identifier).

This study will be conducted according to the principles of the Declaration of Helsinki, version of 2008 and in accordance with the Medical Research Involving Human Subjects Act (WMO, as well as according to the ICH GCP Guideline E6 (1996), EU Directive 2001/20/EC and applicable regulatory requirements and guidelines in the participating countries/regions. Before the first subject has been enrolled in the trial, all ethical and legal requirements were met.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a high level of impulsivity (with or without ADHD) based on a CGI-S-score ≥ 4.
* An Affective Reactivity Index (ARI) score ≥5 indicating a high level of multi dimensional impulsivity.
* Research diagnosis of attention-deficit/hyperactivity disorder (ADHD) and/or borderline personality disorder (BPD) confirmed by structured diagnostic interview according to DSM-5 (ADHD: Diagnostic Interview for Adult ADHD (DIVA 2.0); BPD: Structured Clinical Interview for DSM-IV (SCID-II)).
* Not currently taking any antibiotics or probiotics.
* Deemed reliable and compliant with the protocol by the investigator.
* Ability to speak and comprehend the native language of the country in which the assessments take place.

Exclusion Criteria:

* Subject is being treated with a concomitant medication which is prohibited within this study according to the list of prohibited medications.
* Patients must be on stable medication (i.e. current dose is given since more than 30 days): up-titration is not allowed and careful clinical screening is done at all visits to check whether lower dosage is needed due to increased side effects as a result of treatment with Synbiotic2000Forte.
* Presence of major psychiatric disorders with psychotic's symptoms.
* Neurological disorder involving brain or other central function (e.g., intellectual disability with an assessed IQ < 70, epilepsy, MS, narcolepsy) or other major psychiatric condition requiring hospitalization (e.g., significant mood disorder or psychosis).
* Major physical illness of the cardiovascular, endocrine, pulmonal, or the gastrointestinal system.
* History of or present clinically relevant somatic acute or chronic disorder that, in the opinion of the investigator, might confound the results of tolerability/safety assessment, or prohibit the patients from completing the study, or would not be in the best interest of the patient.
* Subject has a documented allergy, hypersensitivity, or intolerance to any of the ingredients of the intervention.
* Subject has taken another investigational product or taken part in a clinical study within 30 days prior to entering the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Change in the self-rating of affective reactivity (ARI-S) | Assessed at Baseline, at week 5, week 10 and week 11.
Clinical Global Impression - Improvement (CGI-I) total score of 1 or 2 (much improved, very much improved). | assessed at weeks 5, 10, and 11.

SECONDARY OUTCOMES:
Change in Clinical Global Impression - Severity (CGI-S) | Screnning assessment and again at weeks 1, 5 and 10.
Change in ADHD symptom severity total score | Baseline assessment and again at weeks 5, and 10.
  assessed by the Adult Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS). The ADHD-RS is a 18-items scale self-report version for assessing symptoms for ADHD DSM-IV. It consists of a subscale of inattention (IN, 9-items), another of hyperactivity/impulsivity (H / I, 9-items) and the total (TOT, 18-items). The interviewees are asked about the frequency of the symptoms over the past 6 months. Each item is scored from 0 to 3 points, and the highest scores indicates more severe symptomatology of ADHD.
Change in impulsive behaviour | Baseline assessment and again at weeks 5, and 10.
  assessed by the self-rated multi-dimensional impulsivity (UPPS-P)
Change in Self/other rating of aggression and emotional lability (SDQ) | Baseline assessment and again at weeks 5, and 10.
Change in Clinician rating of compulsivity (Y-BOCS) | Baseline assessment and again at weeks 5, and 10.
Change in sleep problems | Baseline assessment and again at weeks 5, and 10.
  5-item questionnaire.
Change in the somatic complaints and side effects describe by the patient. | assessed at weeks 5, 10, and 11.
Change in body composition parameters | Baseline assessment and again at weeks 5, and 10.
  Change in weight in kilograms
Changes in concentrations of blood biomarkers including hormones, neurotransmitters and nutrients. | Baseline assessment and again at weeks 5, and 10.
Change in microbiome composition | Baseline assessment and again at weeks 5, and 10.
Change in nutritional intake | Baseline assessment and again at weeks 5, and 10.
  Participants will be asked to complete at least three 24-h dietary recall (24HDR) per visit, including two week days and one weekend day (non-consecutive days).
Treatment adherence | Baseline assessment and again at weeks 5, and 10.
  Probabilistic Medication Adherence Scale (ProMAS); The total score ranges from 0-18 with a higher score indicating better adherence. Each item is scored as yes (1) or No (0).
Change in functioning problems | Baseline assessment and again at weeks 5, and 10.
  Functioning Assessment Short Test (FAST )
Self-rating of emotion regulation difficulties | Baseline assessment and again at weeks 5, and 10.
  assessed by Difficulties in Emotion Regulation Scale (DERS-16). The total score ranges from 16-80 with a higher score indicating higher difficulties in emotion regulation. Each item is scored as Almost never (1), Somtimes (2), About half the time (3), Most of the time (4), Almost always (5).
Change in gastrointestinal symptoms | Baseline assessment and again at weeks 5, 10, and 11.
  assessed by Bristol Stool Scale;
  There are seven types of stool in the Bristol Stool Scale:
  * Type 1: Separate hard lumps, like nuts (difficult to pass and can be black)
  * Type 2: Sausage-shaped, but lumpy
  * Type 3: Like a sausage but with cracks on its surface (can be black)
  * Type 4: Like a sausage or snake, smooth and soft (average stool)
  * Type 5: Soft blobs with clear cut edges
  * Type 6: Fluffy pieces with ragged edges, a mushy stool (diarrhoea)
  * Type 7: Watery, no solid pieces, entirely liquid (diarrhoea) Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicating lack of dietary fiber, and 6 and 7 indicate diarrhoea.
Change in physical activity: Duration of the activity | Baseline assessment and at week 10.
  parameter measured with a movement sensor.The actigraphy records the duration of the activity. The activity report outcomes how long the participant move (days/hours/min).
Change in physical activity: Intensity of the activity | Baseline assessment and at week 10.
  parameter measured with a movement sensor. The actigraphy records the intensity of the activity. The report of activity outcomes the intensity of the movement classified in four categories from lowest intensity to highest intensity; these categories are:
  * sedentary
  * light
  * moderate
  * vigorous
Change in neurocognitive measure: Detectability | Baseline assessment and again at weeks 5 and 10.
  assessed by Conners' Continuous Performance Test II (CPTII). Assessment duration: 14min.
  Physicological parameter assessed:
  - Detectability (d'): this is a measure of how well the respondent discriminates non-targets (i.e. the letter X) from targets (i.e. all the other letters). This variable is also a signal detection statistic that measures the difference between the signal (targets) and noise (non-targets) distributions. On the Conners CPT-II, d' is reverse scored so that higher raw score and T-score values indicate worse performance (i.e. poorer discrimination)
Change in neurocognitive measure: Omissions | Baseline assessment and again at weeks 5 and 10.
  assessed by Conners' Continuous Performance Test II (CPTII). Assessment duration: 14min.
  Physicological parameter assessed:
  - Omissions (%): Omissions are missed targets. High omissions error rates indicate that the respondent was not responding to the target stimuli due to a specific reason (e.g. difficulty focusing). Omission errors are generally an indicator of inattentiveness.
Change in neurocognitive measure: Commissions | Baseline assessment and again at weeks 5 and 10.
  assessed by Conners' Continuous Performance Test II (CPTII). Assessment duration: 14min.
  Physicological parameter assessed:
  - Commissions (%): Commissions are incorrect responses to non-targets. Depending on the respondent's HRT, high commission error rates may indicate either inattentiveness or impulsivity. If high commission error rates are coupled with slow reaction times, then the respondent was likely inattentive to the stimulus type being presented and thus responded to a high rate of non-targets. If high commission error rates are combined with fast reaction times, the respondent was likely rushing to respond and failed to control his or her impulses when responding to the non-targets. In the latter case, high commission error rates would reflect impulsivity rather than inattentiveness.
Change in neurocognitive measure: Perseverations | Baseline assessment and again at weeks 5 and 10.
  assessed by Conners' Continuous Performance Test II (CPTII). Assessment duration: 14min.
  Physicological parameter assessed:
  - Perseverations (%): Perseverations are responses that are made in less than 100 milliseconds following the presentation of a stimulus. Normal expectations of physiological ability to respond make it virtually impossible for a respondent to perceive and react to a stimulus so quickly. Perseverations are unusually either slow responses to a preceding stimulus, a random response, an anticipatory response, or a repeated response without consideration of the task requirements. Perseverations may be related to impulsivity or an extremely liberal response style. Perseverations are, therefore, likely the result of anticipatory, repetitive, or impulsive responding.
Change in neurocognitive measure: Hit Reaction Time (HRT) | Baseline assessment and again at weeks 5 and 10.
  assessed by Conners' Continuous Performance Test II (CPTII). Assessment duration: 14min.
  Physicological parameter assessed:
  - Hit Reaction Time (HRT): HRT is the mean response speed, measured in milliseconds, for all non-perseverative responses made during the entire administration. An atypically slow HRT may indicate inattentiveness (especially when error rates are high), but it may also be the results of a very conservative response style. Alternatively, a very fast HRT, when combined with high commission error rates, may indicate impulsivity.
Change in neurocognitive measure: Hit Reaction Time Standard Deviation (HRT SD) | Baseline assessment and again at weeks 5 and 10.
  assessed by Conners' Continuous Performance Test II (CPTII). Assessment duration: 14min. .
  Physicological parameter assessed:
  - Hit Reaction Time Standard Deviation (HRT SD): HRT SD measures the consistency of response speed to targets for the entire administration. A high HRT SD indicates greater inconsistency in response speed. Response speed inconsistency is sometimes indicative of an inattentiveness, suggesting that the respondent was less engaged and processed stimuli less efficiently during some parts of the administration.
Change in neurocognitive measure: Variability | Baseline assessment and again at weeks 5 and 10.
  assessed by Conners' Continuous Performance Test II (CPTII). Assessment duration: 14min.
  Physicological parameter assessed:
  - Variability: Variability, like HRT SD, is a measure of response speed consistency, however, Variability is a "within respondent" measure (i.e. the amount of variability the respondent showed in 18 separate sub-blocks of the administration in relation to his or her overall HRT SD score). Although Variability is a different measure than HRT SD, the two measures typically produce comparable results and are both related to inattentiveness. High response speed variability indicates that the respondent's attention and processing efficiency varied throughout the administration.
Change in self-rating of perceived stress. The total score ranges from 0-40 with a higher score indicating higher perceived stress. Each item is scored as Never (0), Almost never (1), Sometimes (2), Fairly Often (3), Very Often (4). | Baseline assessment and at week 10.
  assessed by Perceived Stress Scale (PSS)

CONTACTS AND LOCATIONS:
Locations (3):
- Universitätsklinikum Frankfurt - Goethe Universität, Frankfurt, Germany
- Semmelweis University, Budapest, Hungary
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arteaga-Henriquez G, Ramos-Sayalero C, Ibanez-Jimenez P, Karina Rosales-Ortiz S, Kilencz T, Schiweck C, Schnorr I, Siegl A, Arias-Vasquez A, Bitter I, Fadeuilhe C, Ferrer M, Lavebratt C, Matura S, Reif A, Rethelyi JM, Richarte V, Rommelse N, Antoni Ramos-Quiroga J. Efficacy of a synbiotic in the management of adults with Attention-Deficit and Hyperactivity Disorder and/or Borderline Personality Disorder and high levels of irritability: Results from a multicenter, randomized, placebo-controlled, "basket" trial. Brain Behav Immun. 2024 Aug;120:360-371. doi: 10.1016/j.bbi.2024.06.012. Epub 2024 Jun 15. PMID 38885746
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174
- [Derived] Arteaga-Henriquez G, Rosales-Ortiz SK, Arias-Vasquez A, Bitter I, Ginsberg Y, Ibanez-Jimenez P, Kilencz T, Lavebratt C, Matura S, Reif A, Rethelyi J, Richarte V, Rommelse N, Siegl A, Ramos-Quiroga JA. Treating impulsivity with probiotics in adults (PROBIA): study protocol of a multicenter, double-blind, randomized, placebo-controlled trial. Trials. 2020 Feb 11;21(1):161. doi: 10.1186/s13063-019-4040-x. PMID 32046750